CLINICAL TRIAL: NCT06361511
Title: The Foods & Oil to Repair, Correct and Enhance Strength (FORCES) Study: Determining the Effect of Dietary Oils on Muscle Function, Strength and Mass
Brief Title: The Foods & Oil to Repair, Correct and Enhance Strength (FORCES) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Martha Belury, Professor and Chair, Food Science and Technology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023H0284
Record Dates: First submitted 2024-04-05; First posted 2024-04-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Linoleic Safflower Oil (Experimental): consumption of 12g of high linoleic safflower oil every day
  Interventions: Other: High Linoleic Acid Foods
- High Oleic Safflower Oil (Placebo Comparator): Consumption of 12g of high oleic safflower oil every day
  Interventions: Other: High Oleic Acid Foods

INTERVENTIONS:
Other: High Linoleic Acid Foods — Two food products containing 6g of high linoleic safflower oil each will be consumed each day for a total of 12g daily
  Arms: High Linoleic Safflower Oil
Other: High Oleic Acid Foods — Two food products containing 6g of high oleic safflower oil each will be consumed each day for a total of 12g daily
  Arms: High Oleic Safflower Oil

SUMMARY:
The proposed research is a parallel arm, randomized placebo-controlled clinical trial designed to assess changes in muscle strength, volume, fatigue resistance, and mobility in older adults after daily consumption of 12g of linoleic acid-rich oil.

DETAILED DESCRIPTION:
Study Objectives

1. To assess the effect of linoleic acid supplementation on muscle strength, muscle volume, fatigue- resistance, and physical mobility.
2. To quantify the impact of linoleic acid supplementation on cardiolipin species and mitochondrial function in skeletal muscle of older adults

ELIGIBILITY:
Inclusion Criteria:

* Linoleic Acid Intake <75% of the adequate intake
* Probable sarcopenia

Exclusion Criteria:

* Gastrointestinal diseases or disorders (including pancreatic and gastric bypass surgery) where consumption of the study foods would be contraindication or where the disease or disorder could negatively affect nutrient absorption and/or would prevent participants from tolerating the study foods
* Hyperthyroidism diagnosis
* Food Allergy or intolerances
* Any dietary restriction where consumption of the study foods or any ingredient would be contraindicated
* Unstable management of heart failure, heart disease events (including stroke or heart attack) within last 3 months prior to enrollment, a plan for heart surgeries or cardiac procedures
* Current or previous diagnosis of severe kidney failure, liver cirrhosis, other liver diseases/infections that cause liver damage and some pulmonary diseases or severe/uncontrolled pulmonary diseases
* Severe or uncontrolled rheumatologic or orthopedic diseases
* Current diagnosis of or current treatment of cancer other than non-melanoma skin cancer
* Neuromuscular or neurological conditions or diseases or use of mobility assistance (wheelchair, walker etc..) that would impact movement needed to perform the muscle function tests or prevent completion of the muscle function tests
* Use of mobility assistance (wheelchair, walker etc..) that would prevent completion of the muscle function tests
* Current use of supplements or medications for weight loss or following a weight loss program
* Use of supplements high in linoleic acid in the past 4 weeks prior to enrolling
* Pregnancy and lactation
* Alcohol or drug abuse
* Allergy/intolerance to lidocaine or similar medication
* Use of anticoagulant, antiplatelet, or other blood thinner medications
* Terminal Illness
* Any condition leading to muscle loss or weakness, impaired mobility or range of motion in legs (excluding normal aging)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes is leg extensor muscle strength | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on isokinetic leg extensor muscle strength through isokinetic dynamometer

SECONDARY OUTCOMES:
Changes in quadriceps muscle volume | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on quadriceps muscle volume through MRI
Change in maximum leg press strength | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on maximum leg press strength using leg press machine
Change in leg fatiguability | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on muscle fatiguability through isokinetic dynamometer
Change in muscle mitochondria function | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on muscle and peripheral blood mononuclear cell mitochondria oxygen consumption rate using the Oroboros instrument
Changes in cardiolipin species | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on muscle and peripheral blood mononuclear cell cardiolipin species measured using electrospray ionization-mass spectrometry coupled to high-performance liquid chromatography.
Changes in grip strength | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on grip strength measured using hand dynamometer.
Changes in gait speed | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on gait speed measured by timing a 400-meter walk.
Changes in chair rise time | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on chair rise time measured by timing rise from a seated position five times.
Changes in stair climb power | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on stair climb time measured by timing the completion of climbing 1 flight of stairs
Change in short physical performance battery score | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on short physical performance battery short score which is calculated by measured by measuring time it takes to walk 4 meters, rise from a chair 5 times and the ability to balance in 3 standing positions for 10 seconds each. Scores range from 0 (predicts for worst physical performance) to 12 (predicts for best physical performance)
change in blood fatty acids | Week 0 and Week 24
  To determine the impact of high linoleic safflower oil on changes in blood fatty acids using gas chromatography

OTHER OUTCOMES:
Association of changes in plasma linoleic acid with muscle function | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in plasma linoleic acid with changes in leg extensor muscle strength
Association of changes in plasma linoleic acid with muscle strength | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in plasma linoleic acid with changes in maximum leg press strength
Association of changes in plasma linoleic acid with muscle volume | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in plasma linoleic acid with changes in muscle volume measured by MRI
Association of changes 4-LA-cardiolipin with muscle function | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in 4-LA-cardiolipin with changes in leg extensor muscle strength
Association of changes 4-LA-cardiolipin with muscle strength | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in 4-LA-cardiolipin with changes in maximum leg press strength.
Association of changes 4-LA-cardiolipin with muscle volume | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in 4-LA-cardiolipin with changes in leg muscle volume measured by MRI
Association of changes mitochondria function with muscle volume. | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in mitochondria function with changes in leg muscle volume measured by MRI
Association of changes mitochondria function with muscle function | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in mitochondria function with changes in leg extensor muscle strength.
Association of changes mitochondria function with muscle strength. | Week 0 and Week 24
  Use multiple linear regressions to determine the association of change in mitochondria function with changes in maximum leg press strength.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Belury, PhD RDN, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States